CLINICAL TRIAL: NCT06009835
Title: An Open, Single Center Clinical Study Based on DarwinOncoTreatTM (DOTr) and DarwinOncoTargetTM (DOTa) Algorithm Guidance for Treating Solid Tumor Patients Who Are Exhausted or Unable to Tolerate Standard Treatment Regimens
Brief Title: DOTr/DOTa Algorithm Guidance for Refractory Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DOTr/DOTa for Solid Tumor
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor; Individuation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Treatment group based on DOTr/DOTA detection result: Develop a final treatment plan based on DOTr/DOTA test results, MTB consultation expert opinions, and drug accessibility
  Interventions: Other: Recommended treatment plan

INTERVENTIONS:
Other: Recommended treatment plan — Develop a final treatment plan based on DOTr/DOTA test results, MTB consultation expert opinions, and drug accessibility

SUMMARY:
This study is an open, single center clinical study targeting solid tumor patients who have exhausted or cannot tolerate standard treatment regimens. The main purpose of this study is to investigate the feasibility, efficacy, and safety of selecting treatment regimens based on DOTr/DOTa results for solid tumor patients who have exhausted or cannot tolerate standard treatment regimens.

DETAILED DESCRIPTION:
Both OncoTarget(DarwinOncoTargetTM (DOTa)), which identifies high-affinity inhibitors of individual master regulator (MR) proteins, and OncoTreat(DarwinOncoTreatTM (DOTr)), which identifies drugs that invert the transcriptional activity of hyperconnected MR modules, produced highly significant 30-day disease control rates (68% and 91%, respectively).

ELIGIBILITY:
Inclusion Criteria:

1. The subjects must be able to understand the procedures and methods of this study, be willing to strictly follow the clinical trial protocol to complete this trial, and voluntarily sign a written informed consent form;
2. Patients aged ≥ 18 years old;
3. Solid tumor patients who are depleted of standard treatment or unable to tolerate standard treatment regimens;
4. According to the RECIST solid tumor efficacy evaluation criteria, there should be at least one measurable lesion;
5. ECOG PS score 0-4 (3-4 score only for patients caused by tumor);
6. The expected survival period is not less than 12 weeks;
7. Women of childbearing age must have a Pregnancy test (serum) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the test period and within 8 weeks after the last administration of the test drug;
8. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up;
9. If the main organs function normally, they meet the following standards:

The blood routine examination standard must comply with (no blood transfusion or blood products within 14 days, no correction using G-CSF or other hematopoietic stimulating factors): Hb ≥ 90g/L; ANC ≥ 1.5 × 109/L; PLT ≥ 90 × 109/L;Biochemical examination must meet the following standards: TBIL ≤ 1 × ULN; ALT, AST ≤ 1.5 × ULN; ALP ≤ 2.5 × ULN; BUN and Cr ≤ 1.5 × ULN; Color Doppler echocardiography: left ventricular Ejection fraction (LVEF) ≥ 50%.

Exclusion Criteria:

1. Severe heart disease or discomfort that cannot be treated;
2. Those who suffer from mental illness or abuse of psychotropic substances and are unable to cooperate;
3. Pregnant or lactating female patients;
4. Participating in other clinical trials at the same time;
5. Researchers believe that individuals are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid tumor patients who are exhausted or unable to tolerate standard treatment regimens
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-08-07 (Actual); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of selecting treatment plans based on DOTr/DOTA result | Through study completion, an expected average of 2year
  The proportion of patients who successfully develop treatment plans based on DOTr and DOTa test

SECONDARY OUTCOMES:
ORR | Through study completion, an expected average of 1 year
  Objective response rate (ORR) based on RECIST 1.1 criteria for patients receiving recommended treatment regimens
PFS2/PFS1 | Through study completion, an expected average of 1 year
  he progression free survival (PFS1) after the most recent treatment before enrollment is defined as the progression of the disease from the most recent treatment before enrollment;
  The progression free survival period (PFS2) after enrollment is defined as the time from matched targeted therapy or unmatched therapy to disease progression or death
AEs | Through study completion, an expected average of 1 year
  Number of participants with adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: HaiTao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Mundi PS, Dela Cruz FS, Grunn A, Diolaiti D, Mauguen A, Rainey AR, Guillan K, Siddiquee A, You D, Realubit R, Karan C, Ortiz MV, Douglass EF, Accordino M, Mistretta S, Brogan F, Bruce JN, Caescu CI, Carvajal RD, Crew KD, Decastro G, Heaney M, Henick BS, Hershman DL, Hou JY, Iwamoto FM, Jurcic JG, Kiran RP, Kluger MD, Kreisl T, Lamanna N, Lassman AB, Lim EA, Manji GA, McKhann GM, McKiernan JM, Neugut AI, Olive KP, Rosenblat T, Schwartz GK, Shu CA, Sisti MB, Tergas A, Vattakalam RM, Welch M, Wenske S, Wright JD, Canoll P, Hibshoosh H, Kalinsky K, Aburi M, Sims PA, Alvarez MJ, Kung AL, Califano A. A Transcriptome-Based Precision Oncology Platform for Patient-Therapy Alignment in a Diverse Set of Treatment-Resistant Malignancies. Cancer Discov. 2023 Jun 2;13(6):1386-1407. doi: 10.1158/2159-8290.CD-22-1020. PMID 37061969